CLINICAL TRIAL: NCT07027241
Title: Multicomponent Exercise and Nutrition Based Frailty Intervention in Postoperative Hip Fracture Inpatients
Brief Title: Frailty Intervention in Postoperative Hip Fracture Inpatients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Health Service Executive, Ireland (Other)
Responsible Party: Principal Investigator, Arveen Jeyaseelan, Co-Investigator, Royal College of Surgeons, Ireland
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 24225A007
Record Dates: First submitted 2025-05-29; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Hip Fractures (ICD-10 72.01-72.2); Frailty at Older Adults; Strength Training; Resistance Training; Exercise Training; Protein Supplementation
Keywords: Hip fracture; Exercise; Nutrition; Protein supplementation; Strength and resistance training; Frailty
MeSH Terms: conditions — Hip Fractures; Motor Activity; Frailty | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Study will first be conducted in usual care group and subsequent progress to intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): This arm will assess all aspects of usual postoperative hip fracture care which will include multidisciplinary team assessment which include physiotherapists, occupational therapists, dieticians as well as specialist nurses and doctors working as part of the orthogeriatric team (falls and bone health assessment). They will receive daily physiotherapy training starting on the first postoperative day which will include mobility, balance, strength and gait training. This group will also receive additional protein supplementation in the form of a nutritional supplement twice daily as part of usual postoperative hip fracture care.
  All patients will undergo baseline assessments including assessment of level of frailty, pre-fracture level of mobility & function, postoperative mobility, nutritional status/ screening, grip strength and level of pain.
  All patients will be asked to maintain a three-day food diary to monitor their protein intake.
  Interventions: Other: Usual Care
- Exercise and Nutritional Intervention (Experimental): This arm will include and exercise and nutritional intervention in addition to usual postoperative hip fracture care.
  The exercise program will be delivered 3-5 times per week, each session lasting between 20-30 minutes depending on patient tolerance. The program will be progressed gradually between sessions and be guided by patient tolerance. The program will involve bed/ chair-based aerobic and resistance training (using an arm crank ergometer, resistance bands and ankle weights). The program will be delivered over the entire length of a patient's hospital stay up to a duration of 6 weeks for prolonged stays.
  The nutritional intervention will take the form of a protein fortified evening snack administered by nursing staff (additional 20g of protein).
  All patients will undergo baseline assessments including assessment of level of frailty, pre-fracture level of mobility & function, postoperative mobility, nutritional status/ screening, grip strength and level of pain.
  Interventions: Behavioral: Exercise Intervention; Dietary Supplement: Nutritional Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — This arm will include and exercise and nutritional intervention in addition to usual postoperative hip fracture care.
  The exercise program will be delivered 3-5 times per week, each session lasting between 20-30 minutes depending on patient tolerance. The program will be progressed gradually between sessions and be guided by patient tolerance. The program will involve bed/ chair-based aerobic and resistance training (using an arm crank ergometer, resistance bands and ankle weights). The program will be delivered over the entire length of a patient's hospital stay up to a duration of 6 weeks for prolonged stays.
  All patients will undergo baseline assessments including assessment of level of frailty, pre-fracture level of mobility & function, postoperative mobility, nutritional status/ screening, grip strength and level of pain.
  Other Names: Strength and Resistance Training; Aerobic Training
  Arms: Exercise and Nutritional Intervention
Other: Usual Care — This arm will assess all aspects of usual postoperative hip fracture care which will include multidisciplinary team assessment which include physiotherapists, occupational therapists, dieticians as well as specialist nurses and doctors working as part of the orthogeriatric team (falls and bone health assessment). They will receive daily physiotherapy training starting on the first postoperative day which will include mobility, balance, strength and gait training. This group will also receive additional protein supplementation in the form of a nutritional supplement twice daily as part of usual postoperative hip fracture care.
  All patients will undergo baseline assessments including assessment of level of frailty, pre-fracture level of mobility & function, postoperative mobility, nutritional status/ screening, grip strength and level of pain.
  All patients will be asked to maintain a three-day food diary to monitor their protein intake.
  Other Names: Usual Postoperative Hip Fracture Care
  Arms: Usual Care
Dietary Supplement: Nutritional Intervention — The nutritional intervention will take the form of a protein fortified evening snack administered by nursing staff (additional 20g of protein).
  Other Names: Protein Supplementation
  Arms: Exercise and Nutritional Intervention

SUMMARY:
Hip fracture is a big health concern in older adults, and can lead to increased risk of death, reduced level of independence & mobility, reduced quality of life, and higher likelihood of admission to nursing homes. Frailty is a medical condition associated with ageing that results in a reduced ability to do daily tasks. A frail older adult is also less able to recover well from conditions that may affect their wellbeing (for example, infections, falls resulting in injuries or hospital admissions). Frailty is common in older adults with hip fractures.

There has been increasing research showing that frailty can be slowed down and improved by a combination of nutritional supplementation and exercise. However, most of the research in this area has been in frail older adults living at home or in nursing homes. The exercise or nutritional programs in these studies tend to be carried out over weeks or months. There are very few studies looking at older adults in hospital and how exercise and nutrition help with frailty over shorter periods of time, even more so in patients who have sustained an injury.

There is, however, very little research in hospital based frailty programs in older patients who have suffered major trauma. It is well known that standing up and starting to walk soon after a hip fracture improves time to recovery, reduces hospital length of stay and death. Hence, physiotherapy on the first day after hip fracture surgery is now recommended. However, there needs to be more research to aid in developing physiotherapy and exercise programs that are safe and doable in the care of hip fracture patients despite limited resources in our healthcare system.

Similarly, although malnutrition is common in frail older adults with hip fractures, the benefits of nutritional supplementation in these patients is not fully understood. It is known that having a hip fracture puts a person at risk of muscle breakdown and increasing protein intake is recommended to help reduce this risk. Research on exercise and nutrition based frailty programs specific to hip fracture patients is strongly needed, specifically the development of that are doable and safe in the hospital setting that can help improve outcomes in hip fracture patients after surgery.

The investigators believe that a multicomponent exercise and nutrition based frailty program will be safe, doable and acceptable in frail older adults after hip fracture surgery.

DETAILED DESCRIPTION:
Hip fractures are often the result of falls in the frail older population and result in subsequent poor quality of life and mortality.Over a third of older adults die in the first year after having sustained a hip fracture, suggesting that this may be a result of frailty and the beginning of a decline towards end of life. The incidence of patients presenting with hip fractures is predicted to rise to 11.9% in 2030 compared to 2010. Hip fracture care contributes to a significant burden towards healthcare systems, costing approximately £25,000 per episode and almost £1 billion per annum in the United Kingdom. This likely stems from the likelihood of its association with longer hospital length of stays, multimorbidity and readmissions. Frailty, an age related impairment of physical reserves and resilience, is common in hip fracture patients, and plays a significant role in determining outcomes in this cohort.

Current recommendations suggest early mobilisation post hip fracture to facilitate return to pre-fracture mobility and independence. Intensive in-hospital rehabilitation of post hip fracture patients have been shown to impart greater improvements in physical function and activities of daily living. Hence, physiotherapy on the first day postoperatively is now a recognized quality standard. To supplement this, it is recommended that rehabilitation be provided by multidisciplinary healthcare teams to maximize potential for return to pre-fracture level of function.

The prevalence of malnutrition in hip fracture patients is often high. The management of this problem, particularly in hip fracture patients is challenging. Reduced oral intake in older inpatients are often multifactorial. Studies involving monomodal nutritional interventions in hip fracture patients have shown mixed results. It has been shown that early nutritional intervention led by dieticians was associated with lower prevalence of malnutrition and incidence of pressure ulcers. There was also an association with reduced subacute length of stay. Another study demonstrated that combined nutritional counselling and intensive nutritional intervention led by a dietician reduced malnutrition and improved dietary intake, but only for the duration of the intervention. However, a Cochrane review concluded that nutritional supplementation in the aftercare of hip fracture patients had unclear benefit on outcomes and more randomised trials with robust methodology are required.

There is now an established body of evidence that frailty is modifiable through a combination of nutrition and exercise. However, most of the studies to date have examined interventions delivered over longer periods (e.g. months); and in the community setting. There is however, emerging evidence of in-hospital multicomponent interventions targeting physical and non-physical components of frailty. A recent study showed that a multicomponent intervention in frail and pre-frail adults with cardiovascular disease was safe and feasible in the acute setting. This encompassed additional encouragement to mobilize between usual physiotherapy visits and eat during meals. Additional cognitive stimulation activities and screening and addressing iron deficiency anaemia were also performed bi-daily. It has been shown that an in-hospital multidomain intervention that included nutrition and frailty education and advice, an exercise intervention and cognitive stimulation activities improved frailty and activities of daily living at time of discharge as well as reduced length of stay and subsequent healthcare utilisation.

There is still a relative paucity of research in frailty interventions in older patients who sustained major trauma, and in particular in multi-modal interventions. Studies to date in this population have explored interventions aiming to enhance recovery post-hip fracture for frail patients, however specifically looked at mono-modal interventions, included outpatient interventions in the analyses or only addressed specific components of frailty separately such as cognitive impairment or sarcopenia in the evaluation of rehabilitation strategies in this cohort.

The objective of this study is to assess the feasibility of this intervention in the acute postoperative aftercare of frail older inpatients with hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* Older adults >/= 65
* Clinical Frailty Score 4-6 (This includes patients with very mild, mild and moderate frailty. This would be in keeping with literature quoting frailty interventions where patients who are 'pre-frail' and frail are included)
* Post fragility hip fracture (including subtrochanteric fracture)
* Post hip fracture surgery (all types including total hip replacement, hemiarthroplasty, IM nailing)
* Medically stable postoperatively
* No weightbearing restriction
* Mobile pre-admission (including aids and max assist of 1 person)

Exclusion Criteria:

* Medically unstable (NEWS >3, unless a higher cutoff is stipulated by the primary medical researcher)
* Non fragility hip fracture (fracture from non osteoporotic aetiology, pathologic fracture)
* Hip surgery for other aetiology (prosthetic joint infection, arthritis, implant loosening, avascular necrosis, periprosthetic fracture)
* Polytrauma
* Delirium or severe cognitive impairment (as defined by inability to follow instructions and unable to provide informed consent)
* Pre-existing neurologic or cardiovascular disorders that would affect participation/ compliance with exercise intervention
* Open hip fracture
* Other lower limb orthopaedic disorders that affect participation/ compliance with exercise intervention
* Terminal illness with </= 6 months to live
* Active treatment for cancer (systemic chemotherapy or radiotherapy, patients on oral chemotherapeutic agents/ checkpoint inhibitors will be eligible for inclusion)
* Nursing Home Resident
* Severe lower limb pain post-op
* Severe skin issues/ ulcers in non-operated lower limb that would preclude utilisation of ankle weights
* Swallowing disorders/ difficulty
* Renal impairment with eGFR <30
* Hepatic failure
* Patients with a dairy/ soy allergy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Eligibility Rate | Through study completion, an average of 6 months
  Patients eligible for inclusion/ total number of admissions
Recruitment Rate | Through study completion, an average of 6 months
  Recruited patients/ Patients eligible for inclusion
Number of drop outs | Through study completion, an average fo 6 months
  Number of participant dropouts after recruitment into study
Number of intervention related adverse events | Through study completion, an average of 6 months
  Musculoskeletal injury/ pain, nausea, vomiting, aspiration, constipation etc.
Compliance to prescribed duration of exercise sessions | Through completion of intervention, an average of 3 weeks up to a maximum of 6 weeks
  Percentage of sessions achieving 25 minutes of training
Patient Acceptability of Intervention | Through study completion, an average of 6 months
  Survey utilising open ended questions and 5 point Likert Scales (Strongly Agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree) will be used to evaluate patient satisfaction of the intervention.
Nursing staff acceptability of intervention delivery | Through study completion, an average of 6 months
  Survey utilising open ended questions and 5 point Likert Scales (Strongly Agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree) will be used to evaluate patient satisfaction of the intervention.
Compliance with prescribed intensity | Through completion of intervention, an average of 3 weeks up to a maximum of 6 weeks
  Percentage of sessions completed at Borg Scale score 4-6
Attendance rate | Through completion of intervention, an average of 3 weeks up to a maximum of 6 weeks
  Number of completed sessions/ number of planned sessions
Compliance rate to prescribed nutritional intervention | Through completion of intervention, an average of 3 weeks up to a maximum of 6 weeks
  Number of supplements taken/ number prescribed

SECONDARY OUTCOMES:
Cumulative Ambulation Score (CAS) | At baseline and within 48 hours of discharge from hospital
  Daily score will be 0-6, higher score indicates higher level of independence. Cumulative score over 3 days results in a score of 0-18.
Grip strength (Dominant hand) | At baseline and within 48 hours of discharge from hospital
  Grip strength will be assessed using a handheld dynamometer. Measured in units of kg.
Verbal Rating Scale for Pain (VRS) | At baseline and within 48 hours of discharge from hospital
  Visual scale of 0-3, higher scores indicating more severe pain.
Functional Independence Measure (FIM) | At baseline and within 48 hours of discharge from hospital
  This tool measures activities of daily living, scores range from 18-126, higher scores indicates higher level of independence.
Barthel Index | At baseline and within 48 hours of discharge from hospital
  This tool measures activities of daily living, scored 0-20, higher scores indicates a higher level of independence
Length of Stay (LOS) in hospital | Through intervention completion, an average of 3 weeks up to a maximum of 6 weeks for prolonged stays
  acute hospital stay + super-spell (LOS in acute rehabilitation units)
Discharge Destination | Through intervention completion, an average of 3 weeks up to a maximum of 6 weeks for prolonged stays
  Discharge destination from hospital will be recorded
Health related quality of life (HRQoL) | At baseline and 30 days post discharge
  - Using EuroQol 5-dimension 5-level (EQ-5D-5L) scale. Assesses mobility, self care, activities of daily living, pain, anxiety domains as well as general perception of health. Each dimension on the scale has five response options ranging from no problem to severe problems. The scale also consists of a visual analogue scale, higher values indicate better quality of life.
Upright and Sedentary Events | Throughout inpatient stay, average of 3 weeks up to a maximum of 6 weeks
  Measured using ActivPal Accelerometer
Depression | At baseline and within 48 hours of discharge from hospital
  Screened for using Geriatric Depression Scale (GDS). Screens for depression. Maximum score of 15 points. A score of 5 points or above indicates probable depression.
Fear of Falling | At baseline and within 48 hours of discharge from hospital
  Measured Using the Falls Efficacy Scale- International (FES-I). Scored between 16-64, higher scores indicates increased concern for falling.

CONTACTS AND LOCATIONS:
Overall Officials: Niamh O'Regan, MB BCh BAO, B Med Sci, FRCPI, Principal Investigator — University Hospital Waterford
Locations (1):
- University Hospital Waterford, Waterford, Waterford, Ireland

IPD SHARING:
Plan to Share IPD: No
This will be stored in secure storage for the required duration after completion of study as specified by Good Clinical Practice, after which data will be destroyed.

REFERENCES:
- [Background] Avenell A, Smith TO, Curtain JP, Mak JC, Myint PK. Nutritional supplementation for hip fracture aftercare in older people. Cochrane Database Syst Rev. 2016 Nov 30;11(11):CD001880. doi: 10.1002/14651858.CD001880.pub6. PMID 27898998
- [Background] Saunders J, Smith T. Malnutrition: causes and consequences. Clin Med (Lond). 2010 Dec;10(6):624-7. doi: 10.7861/clinmedicine.10-6-624. No abstract available. PMID 21413492
- [Background] Malafarina V, Reginster JY, Cabrerizo S, Bruyere O, Kanis JA, Martinez JA, Zulet MA. Nutritional Status and Nutritional Treatment Are Related to Outcomes and Mortality in Older Adults with Hip Fracture. Nutrients. 2018 Apr 30;10(5):555. doi: 10.3390/nu10050555. PMID 29710860
- [Background] Audit NOoC. Irish Hip Fracture Database National Report 2023. 2024.
- [Background] Ftouh S, Morga A, Swift C; Guideline Development Group. Management of hip fracture in adults: summary of NICE guidance. BMJ. 2011 Jun 21;342:d3304. doi: 10.1136/bmj.d3304. No abstract available. PMID 21693526
- [Background] Oberstar JS, Bakker CJ, Sorich M, McCarthy T. What Postoperative Nutritional Interventions Lead to Better Outcomes in Fragility Hip Fractures? A Systematic Review. Geriatr Orthop Surg Rehabil. 2023 Feb 15;14:21514593231155828. doi: 10.1177/21514593231155828. eCollection 2023. PMID 36817328
- [Background] Phang JK, Lim ZY, Yee WQ, Tan CYF, Kwan YH, Low LL. Post-surgery interventions for hip fracture: a systematic review of randomized controlled trials. BMC Musculoskelet Disord. 2023 May 25;24(1):417. doi: 10.1186/s12891-023-06512-9. PMID 37231406
- [Background] Cadel L, Kuluski K, Wodchis WP, Thavorn K, Guilcher SJT. Rehabilitation interventions for persons with hip fracture and cognitive impairment: A scoping review. PLoS One. 2022 Aug 15;17(8):e0273038. doi: 10.1371/journal.pone.0273038. eCollection 2022. PMID 35969624
- [Background] Avola M, Mangano GRA, Testa G, Mangano S, Vescio A, Pavone V, Vecchio M. Rehabilitation Strategies for Patients with Femoral Neck Fractures in Sarcopenia: A Narrative Review. J Clin Med. 2020 Sep 26;9(10):3115. doi: 10.3390/jcm9103115. PMID 32993140
- [Background] Halter M, Jarman H, Moss P, Kulnik ST, Baramova D, Gavalova L, Cole E, Crouch R, Baxter M. Configurations and outcomes of acute hospital care for frail and older patients with moderate to major trauma: a systematic review. BMJ Open. 2023 Feb 21;13(2):e066329. doi: 10.1136/bmjopen-2022-066329. PMID 36810176
- [Background] Wang YC, Liang CK, Chou MH, Chiu CF, Lin HC, Hsu YH, Liao MC, Yin CH, Chou MY, Lin YT. The Effectiveness of Frailty Intervention for Older Patients with Frailty during Hospitalization. J Nutr Health Aging. 2023;27(6):413-420. doi: 10.1007/s12603-023-1924-y. PMID 37357324
- [Background] Puts MTE, Toubasi S, Andrew MK, Ashe MC, Ploeg J, Atkinson E, Ayala AP, Roy A, Rodriguez Monforte M, Bergman H, McGilton K. Interventions to prevent or reduce the level of frailty in community-dwelling older adults: a scoping review of the literature and international policies. Age Ageing. 2017 May 1;46(3):383-392. doi: 10.1093/ageing/afw247. PMID 28064173
- [Background] Dedeyne L, Deschodt M, Verschueren S, Tournoy J, Gielen E. Effects of multi-domain interventions in (pre)frail elderly on frailty, functional, and cognitive status: a systematic review. Clin Interv Aging. 2017 May 24;12:873-896. doi: 10.2147/CIA.S130794. eCollection 2017. PMID 28579766
- [Background] Kidd T, Mold F, Jones C, Ream E, Grosvenor W, Sund-Levander M, Tingstrom P, Carey N. What are the most effective interventions to improve physical performance in pre-frail and frail adults? A systematic review of randomised control trials. BMC Geriatr. 2019 Jul 11;19(1):184. doi: 10.1186/s12877-019-1196-x. PMID 31291884
- [Background] Travers J, Romero-Ortuno R, Bailey J, Cooney MT. Delaying and reversing frailty: a systematic review of primary care interventions. Br J Gen Pract. 2019 Jan;69(678):e61-e69. doi: 10.3399/bjgp18X700241. Epub 2018 Dec 3. PMID 30510094
- [Background] Gardner B, Jovicic A, Belk C, Kharicha K, Iliffe S, Manthorpe J, Goodman C, Drennan VM, Walters K. Specifying the content of home-based health behaviour change interventions for older people with frailty or at risk of frailty: an exploratory systematic review. BMJ Open. 2017 Feb 9;7(2):e014127. doi: 10.1136/bmjopen-2016-014127. PMID 28183809
- [Background] Nascimento CM, Ingles M, Salvador-Pascual A, Cominetti MR, Gomez-Cabrera MC, Vina J. Sarcopenia, frailty and their prevention by exercise. Free Radic Biol Med. 2019 Feb 20;132:42-49. doi: 10.1016/j.freeradbiomed.2018.08.035. Epub 2018 Aug 31. PMID 30176345
- [Background] Dong X, Zhang X, Hu F, Yang S, Hong Z, Geng Q. Association of frailty with adverse outcomes in surgically treated geriatric patients with hip fracture: A meta-analysis and trial sequential analysis. PLoS One. 2024 Jun 21;19(6):e0305706. doi: 10.1371/journal.pone.0305706. eCollection 2024. PMID 38905251
- [Background] Song Y, Wu Z, Huo H, Zhao P. The Impact of Frailty on Adverse Outcomes in Geriatric Hip Fracture Patients: A Systematic Review and Meta-Analysis. Front Public Health. 2022 Jun 30;10:890652. doi: 10.3389/fpubh.2022.890652. eCollection 2022. PMID 35844855
- [Background] Forssten MP, Cao Y, Trivedi DJ, Ekestubbe L, Borg T, Bass GA, Mohammad Ismail A, Mohseni S. Developing and validating a scoring system for measuring frailty in patients with hip fracture: a novel model for predicting short-term postoperative mortality. Trauma Surg Acute Care Open. 2022 Sep 13;7(1):e000962. doi: 10.1136/tsaco-2022-000962. eCollection 2022. PMID 36117728
- [Background] Pollock FH, Bethea A, Samanta D, Modak A, Maurer JP, Chumbe JT. Readmission within 30 days of discharge after hip fracture care. Orthopedics. 2015 Jan;38(1):e7-13. doi: 10.3928/01477447-20150105-53. PMID 25611424
- [Background] White SM, Griffiths R, Holloway J, Shannon A. Anaesthesia for proximal femoral fracture in the UK: first report from the NHS Hip Fracture Anaesthesia Network. Anaesthesia. 2010 Mar;65(3):243-8. doi: 10.1111/j.1365-2044.2009.06208.x. Epub 2009 Dec 18. PMID 20039864
- [Background] Maxwell L, White S. Anaesthetic management of patients with hip fractures: an update. Continuing Education in Anaesthesia, Critical Care & Pain. 2013;13(5):179-83.
- [Background] Leal J, Gray AM, Prieto-Alhambra D, Arden NK, Cooper C, Javaid MK, Judge A; REFReSH study group. Impact of hip fracture on hospital care costs: a population-based study. Osteoporos Int. 2016 Feb;27(2):549-58. doi: 10.1007/s00198-015-3277-9. Epub 2015 Aug 19. PMID 26286626
- [Background] Williamson S, Landeiro F, McConnell T, Fulford-Smith L, Javaid MK, Judge A, Leal J. Costs of fragility hip fractures globally: a systematic review and meta-regression analysis. Osteoporos Int. 2017 Oct;28(10):2791-2800. doi: 10.1007/s00198-017-4153-6. Epub 2017 Jul 26. PMID 28748387
- [Background] Stevens JA, Rudd RA. The impact of decreasing U.S. hip fracture rates on future hip fracture estimates. Osteoporos Int. 2013 Oct;24(10):2725-8. doi: 10.1007/s00198-013-2375-9. Epub 2013 Apr 30. PMID 23632827
- [Background] Han CY, Crotty M, Thomas S, Cameron ID, Whitehead C, Kurrle S, Mackintosh S, Miller M. Effect of Individual Nutrition Therapy and Exercise Regime on Gait Speed, Physical Function, Strength and Balance, Body Composition, Energy and Protein, in Injured, Vulnerable Elderly: A Multisite Randomized Controlled Trial (INTERACTIVE). Nutrients. 2021 Sep 13;13(9):3182. doi: 10.3390/nu13093182. PMID 34579060
- [Background] Panula J, Pihlajamaki H, Mattila VM, Jaatinen P, Vahlberg T, Aarnio P, Kivela SL. Mortality and cause of death in hip fracture patients aged 65 or older: a population-based study. BMC Musculoskelet Disord. 2011 May 20;12:105. doi: 10.1186/1471-2474-12-105. PMID 21599967
- [Background] Hu F, Jiang C, Shen J, Tang P, Wang Y. Preoperative predictors for mortality following hip fracture surgery: a systematic review and meta-analysis. Injury. 2012 Jun;43(6):676-85. doi: 10.1016/j.injury.2011.05.017. Epub 2011 Jun 17. PMID 21683355
- [Background] Lin HS, Watts JN, Peel NM, Hubbard RE. Frailty and post-operative outcomes in older surgical patients: a systematic review. BMC Geriatr. 2016 Aug 31;16(1):157. doi: 10.1186/s12877-016-0329-8. PMID 27580947
- [Background] van de Ree CLP, Landers MJF, Kruithof N, de Munter L, Slaets JPJ, Gosens T, de Jongh MAC. Effect of frailty on quality of life in elderly patients after hip fracture: a longitudinal study. BMJ Open. 2019 Jul 18;9(7):e025941. doi: 10.1136/bmjopen-2018-025941. PMID 31324679
- [Background] Fountotos R, Ahmad F, Bharaj N, Munir H, Marsala J, Rudski LG, Goldfarb M, Afilalo J. Multicomponent intervention for frail and pre-frail older adults with acute cardiovascular conditions: The TARGET-EFT randomized clinical trial. J Am Geriatr Soc. 2023 May;71(5):1406-1415. doi: 10.1111/jgs.18228. Epub 2023 Jan 16. PMID 36645227